CLINICAL TRIAL: NCT03418623
Title: Effect of GET73 on Magnetic Resonance Spectroscopy Measures of Central Glutamate and GABA and Alcohol Cue-elicited Brain Activation in Recently Abstinent Non-treatment Seeking Individuals With Alcohol Use Disorder.
Brief Title: Effect of GET73 on MRS Measures of Central Glutamate and GABA in Individuals With Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorio Farmaceutico Ct S.r.l. (Industry)
Collaborators: Latis S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GET73 ¹H-MRS
Record Dates: First submitted 2018-01-08; First posted 2018-02-01 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Alcohol Use Disorder
Keywords: Glutamate; Alcohol use; GABA; GET73; Non-treatment seeking
MeSH Terms: conditions — Alcoholism; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: After the eligibility of a subject has been determined in an initial screening period, the study will be conducted in 2 consecutive phases: in the first phase (phase A) the participant will be administered GET73 or placebo in a randomized order, in the other phase (phase B), the participant will be administered the treatment not received during phase A.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be double-blinded. At initiation visit the Investigator will be instructed on the method for blind breaking. The Contract Research Organization (CRO) will provide the Investigator with a set of sealed envelopes, each containing the unblinding information for a patient kit; the envelopes will be kept in the Pharmacy until the end of the study. A second set of sealed envelopes will be kept by the Sponsor pharmacovigilance officer.
  Unblinding codes should only be used in emergency situations for reasons of patient safety. The Investigator should contact the Sponsor before breaking the blind or the Sponsor should be informed immediately afterwards. The reason for breaking the blind must be fully documented and entered on the case report form.
  The unblinding envelopes will be checked for integrity by the Clinical Research Associate (CRA) and returned to the Sponsor at the end of the study.
  The subjects for whom the blind will be broken will be withdrawn from the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GET73 (Experimental): GET73 is administered at the dose of 300 mg t.i.d. per day, with a minimum gap of 4 hours between administrations and a maximum gap of 9 hours. Each subject ingests a total of 5 capsules of GET73: 3 capsules of GET73 on the first day of the related phase, according to randomization, and 2 capsules on the second day of each phase.
  Interventions: Drug: GET73
- Placebo (Placebo Comparator): Placebo is administered t.i.d. per day, with a minimum gap of 4 hours between administrations and a maximum gap of 9 hours. Each subject ingests a total of 5 capsules of Placebo: 3 capsules of Placebo on the first day of the related phase, according to randomization, and 2 capsules on the second day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GET73 — GET73 300 mg oral capsules, administered three times a day on Visit 2 and 4, and twice a day on Visit 3 and 5.
  Arms: GET73
Other: Placebo — Placebo oral capsules, administered three times a day on Visit 2 and 4, and twice a day on Visit 3 and 5.
  Arms: Placebo

SUMMARY:
This study is aimed at examining whether GET73 modulates the indices of central glutamate and γ-aminobutyric acid (GABA) levels in recently abstinent subjects that meet Alcohol Use Disorder (AUD) criteria, as measured by proton nuclear magnetic resonance spectroscopy (¹H-MRS), in order to provide a human translation of the findings demonstrated in different preclinical models, both in vitro and in vivo. In addition, the study will examine the effects of GET73 on alcohol cue induced brain activation by using a well-established blood-oxygen-level-dependent (BOLD) functional magnetic resonance (fMRI) paradigm in the same individuals. In summary, the study should provide important information on (i) the potential mechanism of action of GET73, (ii) on the brain mechanisms that would support its potential use for reduction in craving and drinking in AUD patients, and (iii) expand data on its safe use as a medication in heavy drinking individuals.

DETAILED DESCRIPTION:
This study is aimed at examining whether GET73 modulates the indices of central glutamate and γ-aminobutyric acid (GABA) levels in recently abstinent subjects that meet Alcohol Use Disorder (AUD) criteria, as measured by proton nuclear magnetic resonance spectroscopy (¹H-MRS), in order to provide a human translation of the findings demonstrated in different preclinical models, both in vitro and in vivo. In addition, the study will examine the effects of GET73 on alcohol cue induced brain activation by using a well-established blood-oxygen-level-dependent (BOLD) functional magnetic resonance (fMRI) paradigm in the same individuals. In summary, the study should provide important information on (i) the potential mechanism of action of GET73, (ii) on the brain mechanisms that would support its potential use for reduction in craving and drinking in AUD patients, and (iii) expand data on its safe use as a medication in heavy drinking individuals.

The enrolment period will last approximately 18 to 21 months. For each subject the study will last 25 to 45 days.

The primary objective of the study is to evaluate whether GET73 modulates central glutamate levels in recently abstinent individuals with AUD, using proton nuclear magnetic resonance spectroscopy (¹H-MRS).

The secondary objectives of the study are:

1. To evaluate whether GET73 modulates central GABA levels in recently abstinent individuals with AUD, using proton nuclear magnetic resonance spectroscopy (¹H-MRS)
2. To evaluate whether GET73 affects alcohol cue induced brain activity in reward areas of brain.
3. To explore whether the effects of GET73 on glutamate and GABA levels are related to its effects on alcohol cue induced brain activity.

Safety Objective To evaluate the safety profile of GET73 in individuals with AUD, comparing Adverse Events (AEs) occurrence during GET73 treatment period vs placebo treatment period.

This is a within-subject cross-over, randomized, double-blind, placebo-controlled study.

Being a double blinded study, GET73 and placebo will be packaged identically. Both the Investigator and the study participant will be unaware of the treatment administered.

The investigational product will be supplied to the Center packaged in "patient kits". Each "patient kit" will be made of 2 bottles (bottle A and bottle B) each containing 20 capsules of either GET73 or placebo.

Being a cross-over design, all participants will receive both placebo and active treatment. The sequential order in which they will be administered to each participant will be defined by the randomization list. The participant will always receive bottle A in the phase A of the study and bottle B in phase B, but the content of the two bottles varies according to the randomization list. Research personnel will be blind to the content of the bottles, i.e. what study medication the subject is taking.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants, or females who are post-menopausal or surgically sterile.
2. Age between 21 and 40 years old (inclusive).
3. Meets Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for current Alcohol Use Disorder, moderate severity (4 or more criteria met) as indicated by the Structured Clinical Interview for DSM-5 (SCID-5-RV).
4. Reports drinking, on average, > 20 standard drinks per week in the 90 days prior to screening evaluation, and in the last week prior to screening.
5. Must report drinking within the 48 hours prior to the first dose of medication in each study medication period.
6. Positive for Ethyl Glucuronide (EtG) in urine (> 100 ng/ml) at screening and prior to the first dose of medication in each study medication period.
7. Currently not engaged in, and does not want treatment for, alcohol related problems.
8. Able to read and understand questionnaires and informed consent.

Exclusion Criteria:

1. Current DSM-5 diagnosis of any other substance use disorder except Nicotine Use Disorder.
2. Any psychoactive substance use (except marijuana and nicotine) within the last 30 days before the screening visit, as indicated by self-report and/or urine drug screen.
3. No marijuana use within the last seven days before the screening visit, by verbal report and negative urine drug test (< 50 ng/mL); if positive at screening, must be negative or decreasing urine Delta9-Tetrahydrocannabinol (THC) levels (corrected for urine creatinine level) at the second test (Day1 A-1).
4. Current DSM-5 Axis I diagnosis, including major depression, panic disorder, obsessive-compulsive disorder, post-traumatic stress disorder, bipolar affective disorder, schizophrenia, dissociative disorders, eating disorders, or any other psychotic or organic mental disorder.
5. Current suicidal or homicidal ideation.
6. Need for maintenance or acute treatment with any psychoactive medication, including antiepileptic medications.
7. Current use, or use in the past 30 days, of any medication known to affect alcohol intake (e.g., disulfiram, naltrexone, acamprosate, topiramate).
8. History of severe alcohol withdrawal (e.g., seizure, delirium tremens), as evidenced by self-report or a Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar) score > 10.
9. Clinically significant medical problems (e.g., unstable hypertension, neurological, cardiovascular, renal, gastrointestinal, or endocrine problems) that would impair participation or limit medication ingestion.
10. Current or past hepatocellular disease, as indicated by verbal report or elevations of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 300% the upper limit of the normal range, or bilirubin > 150% the upper limit of the normal range.
11. Lack of a stable living situation.
12. Presence of ferrous metal in the body, as evidenced by metal screening and self-report.
13. Severe claustrophobia or weight > 300 pounds that preclude placement in the MRI scanner.
14. History of head injury with > 2 minutes of unconsciousness.
15. Participation in any behavioral and/or pharmacological study within the past 30 days;
16. Concomitant use of CYP2C19 substrates; use of CYP2C19 and CYP3A4 inhibitors or inducers in the 14 days before dosing.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Concentrations of glutamate in dorsal anterior cingulate measured via Proton Magnetic Resonance Spectroscopy | After 5 doses of medication administered over 2 days, repeated after a wash-out period of 7 to 21 days (crossover design)
  The presence of water and glutamate will be quantified through ¹H-MRS and the change in glutamate/water concentration between baseline and end of treatment will be assessed

SECONDARY OUTCOMES:
Concentrations of GABA in dorsal anterior cingulate measured via Proton Magnetic Resonance Spectroscopy | After 5 doses of medication administered over 2 days, repeated after a wash-out period of 7 to 21 days (crossover design)
  The presence of water and GABA will be quantified through ¹H-MRS and the change in GABA/water concentration between baseline and end of treatment will be assessed
Change in the blood oxygenation level dependent (BOLD) signal to alcohol cues | After 5 doses of medication administered over 2 days, repeated after a wash-out period of 7 to 21 days (crossover design)
  Magnitude of change in the blood oxygenation level dependent (BOLD) signal to alcohol cues, relative to neutral beverage cues, in the ventral striatum and dorsal anterior cingulate cortex (alcohol cue reactivity task described in Schacht et al., 2013)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond F Anton, MD, Principal Investigator — Department of Psychiatry and Behavioral Sciences - Medical University of South Carolina
Locations (1):
- Department of Psychiatry and Behavioral Sciences - Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Schacht JP, Anton RF, Voronin KE, Randall PK, Li X, Henderson S, Myrick H. Interacting effects of naltrexone and OPRM1 and DAT1 variation on the neural response to alcohol cues. Neuropsychopharmacology. 2013 Feb;38(3):414-22. doi: 10.1038/npp.2012.195. Epub 2012 Oct 3. PMID 23032071